CLINICAL TRIAL: NCT07104240
Title: TweenVax: A Comprehensive Practice-, Provider-, and Parent/Patient-Level Intervention to Improve Adolescent HPV Vaccination
Brief Title: A Vaccine Promotion Package (TweenVax) to Improve Adolescent HPV Vaccination, TweenVax Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Robert Bednarczyk, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00009250; NCI-2025-03575 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00009250 (Other: Emory University Hospital/Winship Cancer Institute); RSPH6573-25 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH); R37CA234119 (NIH)
Record Dates: First submitted 2025-07-18; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Human Papillomavirus-Related Carcinoma
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Early Intervention, Educational; Educational Status; Methods; Health Promotion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm I (TweenVax, practice, provider, parent, patient level) (Experimental): Practices receive all TweenVax components and trainings related to the practice, provider and staff, parent and adolescent-level intervention. Parents receive access to the TweenVax application and receive TweenVax vaccination information using the provided tablet during clinical encounters on study.
  Interventions: Other: Educational Intervention; Other: Health Promotion and Education; Other: Internet-Based Intervention
- Arm II (practice and provider) (Experimental): Practices receive components and trainings related to the practice and provider-level intervention on study.
  Interventions: Other: Health Promotion and Education
- Arm III (control) (Active Comparator): Practices continue to offer standard of care adolescent vaccination promotion practices to adolescent patients on study.
  Interventions: Other: Best Practice

INTERVENTIONS:
Other: Best Practice — Offer standard of care adolescent vaccination promotion practices
  Other Names: standard of care; standard therapy
  Arms: Arm III (control)
Other: Educational Intervention — Receive vaccination information
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm I (TweenVax, practice, provider, parent, patient level)
Other: Health Promotion and Education — Receive all TweenVax components and trainings for the practice, providers and staff, parents and adolescents
  Arms: Arm I (TweenVax, practice, provider, parent, patient level)
Other: Health Promotion and Education — Receive components and trainings for the practice and provider levels
  Arms: Arm II (practice and provider)
Other: Internet-Based Intervention — Receive access to TweenVax application
  Arms: Arm I (TweenVax, practice, provider, parent, patient level)

SUMMARY:
This clinical trial compares the effect of a vaccine promotional intervention, TweenVax, to standard of care vaccination promotion practices on rates of human papillomavirus (HPV) vaccination in adolescents. HPV vaccination has been identified as a priority for cancer prevention and control by the Cancer Moonshot Blue Ribbon Panel, which estimated that increasing HPV vaccination rates can prevent 400,000 HPV-related cancers in the next 5-10 years. The goal is for HPV vaccinations to be completed by the age of 13. It has been estimated that only about 16% of adolescents were fully up to date with HPV vaccines by age 13. Strong and consistent provider recommendations have been shown to play an important role in the uptake of vaccines. In addition, education and information received by parents may improve the strength of recommendations by providers. The TweenVax intervention includes practice, provider, parent and patient level education to teach best practices, help with vaccine messaging, and give correct and easy to understand information to parents. Providing practice, provider and parent level access to TweenVax may be more effective than current vaccine promotion practices in improving HPV vaccination rates in adolescents.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To test the expanded and revised TweenVax intervention package based on pilot study findings and formative research evaluating best practices and deficiencies observed during adolescent healthcare encounters.

OUTLINE: Pediatric practices are randomized to 1 of 3 arms.

ARM I: Practices receive all TweenVax components and trainings related to the practice, provider and staff, parent and adolescent-level intervention. Parents receive access to the TweenVax application and receive TweenVax vaccination information using the provided tablet during clinical encounters on study.

ARM II: Practices receive components and trainings related to the practice and provider-level intervention on study.

ARM III: Practices continue to offer standard of care adolescent vaccination promotion practices to adolescent patients on study.

After completion of study intervention, practices are followed for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* PRACTICE-LEVEL: Must be community based primary care providers (pediatrics or family practice)
* PRACTICE-LEVEL: Are willing to be part of the study
* PRACTICE-LEVEL: Have sufficient patient population to support 51 adolescents aged 9-12 years over approximately a 9-month period
* PRACTICE-LEVEL: Utilize an electronic medical records system and/or report to the state Immunization Information System (IIS)
* CHILD/ADOLESCENT: Aged 9-12 years
* CHILD/ADOLESCENT: Seeking care from an enrolled practice during the study period
* CHILD/ADOLESCENT: Have not received any doses of HPV vaccine by the time of their first visit during the study period

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1836 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2027-03-06 (Estimated); Study Completion 2028-03-06 (Estimated)

PRIMARY OUTCOMES:
Initiation and completion of human papillomavirus (HPV) vaccine by 13 years of age | Up to 1 year follow-up
  Will do a direct comparison of rates in the intervention groups relative to the control group. However, if there is an imbalance in covariates between the arms, will then use multivariable regression, accounting for clinic-level clustering and key covariates. If needed, the initial regression model will be a log-binomial regression, to directly estimate relative risk; however, the final modeling choice will be dependent on the actual distribution of the data which may necessitate an alternative modeling method. Each intervention arm will be compared to the control arm independently, and analysis will be conducted separately for HPV vaccine series initiation and completion. Will model vaccination rates with associated 95% confidence intervals, and comparisons between intervention arms will be conducted by comparing confidence intervals.

SECONDARY OUTCOMES:
Rate of missed opportunities for vaccination | Up to 1 year follow-up
  Will assess the total number of healthcare encounters, classifying them as whether the adolescent was eligible for HPV vaccine at the time of the visit. Eligible visits with no vaccine administered, when a vaccine could have been administered based on eligibility, will be considered a missed opportunity. Will compare the mean number of missed opportunities per arm using analysis of variance, and the proportion of adolescents with at least one missed opportunity per arm using Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bednarczyk, PhD, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States